CLINICAL TRIAL: NCT05254171
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Nab-Paclitaxel and Gemcitabine With or Without SBP-101 in Subjects Previously Untreated for Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of Nab-Paclitaxel and Gemcitabine With or Without SBP-101 in Pancreatic Cancer
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Panbela Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-SBP-101-04
Record Dates: First submitted 2022-01-13; First posted 2022-02-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Stage IV
Keywords: SBP-101
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to Experimental Arm vs. Control Arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): SBP-101 + Nab-paclitaxel and Gemcitabine
  Interventions: Drug: SBP-101; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Control Arm (Placebo Comparator): Placebo + Nab-Paclitaxel and Gemcitabine
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Other: Placebo

INTERVENTIONS:
Drug: SBP-101 — small molecule polyamine metabolic inhibitor for subcutaneous injection
  Other Names: ivospemin
  Arms: Experimental Arm
Drug: Nab-paclitaxel — paclitaxel protein-bound particles for injectable suspension
  Other Names: Abraxane
Drug: Gemcitabine — gemcitabine for injection
  Other Names: Gemzar
Other: Placebo — Normal Saline
  Arms: Control Arm

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, multicenter study of standard treatment with nab-paclitaxel and gemcitabine with or without SBP-101 in subjects previously untreated for metastatic pancreatic ductal adenocarcinoma (PDA), including subjects who have received prior neoadjuvant or adjuvant treatment.

DETAILED DESCRIPTION:
This trial will enroll approximately 600 patients to evaluate the effect of SBP-101 on Overall Survival when administered with gemcitabine and nab-paclitaxel compared to gemcitabine and nab-paclitaxel and a placebo. Secondary endpoints include Progression-free survival, radiologic responses to treatment, and Quality of Life measures. An independent, external Data Safety Monitoring Board (DSMB) will monitor safety and efficacy and a planned futility analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
* Is previously untreated for metastatic pancreatic ductal adenocarcinoma; metastatic disease must have been diagnosed within the past 3 months; and subject is expected to receive standard treatment with gemcitabine and nab-paclitaxel. Subjects who have had planned or prior surgery, such as a Whipple procedure, with or without neo-adjuvant/or adjuvant chemotherapy may be included.
* Life expectancy ≥ 3 months.
* Measurable disease on computed tomography (CT) or magnetic resonance imaging (MRI) scan by RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Adult, age ≥ 18 years, male or female.
* Females of child-bearing potential must have a negative serum pregnancy test within 14 days prior to start of study treatment and must use an adequate method of contraception from 2 weeks before the first administration of SBP-101 until 6 months after the last administration of study drug (i.e., last dose of any of the three drugs in the regimen). Female subjects are considered to be of childbearing potential unless they are postmenopausal (at least 12 months of consecutive amenorrhea, without other known or suspected cause) and over 55 years old or have been sterilized surgically (i.e., bilateral tubal ligation, hysterectomy, or bilateral oophorectomy, all with surgery at least one month before dosing).
* Adequate bone marrow, hepatic and renal function as outlined in protocol.
* QTc interval ≤ 470 ms (for women) and ≤ 450 ms (for men) on the ECG at baseline calculated by either the Fridericia or Framingham formula.
* Willing and able to provide written informed consent: voluntary agreement to participate in the study following disclosure of risks and procedures required.

Exclusion Criteria:

* When results of germline or somatic testing done prior to screening are known, subjects known to have mutations of the BRCA 1/2 (Breast Cancer gene) are excluded.
* Concomitant metformin administration. Diabetic subjects on treatment with metformin, or any other derivative thereof, must discontinue it at least 5 days prior to C1D1 and not take metformin while on study (other diabetic medications are allowed).
* Any history of retinopathy or at risk for retinal detachment (personal or family history of retinal detachment, extreme myopia [-6.0 diopters or approximately 20/500], eye surgery <6 months prior to C1D1, or history of a severe eye injury. Subjects with findings of retinopathy on baseline ophthalmology exams will be excluded.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the opinion of the Investigator or Medical Monitor, makes it undesirable for the subject to participate in the study or that would jeopardize compliance with the protocol. Subjects with pre-existing well-controlled diabetes are not excluded.
* Medical or psychiatric conditions that compromise the subject's ability to give informed consent or to complete the protocol or a history of non-compliance.
* Presence of islet-cell or pancreatic neuroendocrine tumor or mixed adenocarcinoma-neuroendocrine carcinoma.
* Symptomatic central nervous system (CNS) malignancy or metastasis. Screening of asymptomatic subjects without history of CNS metastases is not required.
* Serum albumin < 30 g/L (3.0 g/dL).
* Deep vein thrombosis (DVT) or portal vein occlusion, pulmonary embolism (PE), or other thromboembolic event that occurs during screening.
* Presence of known active bacterial, fungal, or viral infection requiring systemic therapy.
* Known active infection with human immunodeficiency virus (HIV), hepatitis B or C.
* Presence of interstitial lung disease, pulmonary fibrosis, or pulmonary hypersensitivity reaction.
* Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV.
* Pregnant or lactating.
* Major surgery within 4 weeks prior to the start of study drug treatment, without complete recovery.
* Known hypersensitivity to any component of study treatments.
* Participation in any other clinical investigation within 4 weeks of receiving the first dose of study drug.
* Any history of hydroxychloroquine use (Plaquenil® and other brand names).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of first dose up to 100 weeks or until death
  Compare OS between subjects who receive SBP-101 and those who do not receive SBP-101 (i.e., placebo) in combination with nab-paclitaxel and gemcitabine

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of first dose up to 100 weeks or until death
  Compare PFS between SBP-101 and placebo

OTHER OUTCOMES:
Overall Objective Response (ORR) | Up to 100 weeks
  Compare ORR between SBP-101 and placebo
Disease Control Rate (DCR) | Up to 100 weeks
  Compare DCR between SBP-101 and placebo
Duration of Response (DoR) | Up to 100 weeks
  Compare DoR between SBP-101 and placebo
Quality of Life (QOL) Questionnaires: EORTC QLC-C30 | Up to 100 weeks
  Compare QOL changes in scores between SBP-101 and placebo
Quality of Life (QOL) Questionnaires: QLQ-PAN26 | Up to 100 weeks
  Compare QOL changes in scores between SBP-101 and placebo
Number of Subjects with treatment-emergent adverse events as assessed by CTCAE v5.0 | Up to 100 weeks
  Compare Safety and Tolerability of SBP-101 to placebo when administered in combination with nab-paclitaxel and gemcitabine
Exploratory | Up to 100 weeks
  Compare effects of SBP-101 and placebo on blood levels of carbohydrate antigen (CA) CA 19-9 and circulating tumor DNA (cT DNA).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Walker, MD, Study Director — Panbela Therapeutics, Inc.
Locations (92):
- United States (14):
  - Genesis Cancer and Blood Institute (SCRI), Hot Springs, Arkansas
  - Providence Medical Foundation, Fullerton, California
  - Yale Cancer Center, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Henry Ford Health System, Detroit, Michigan
  - CentraCare Health, Saint Cloud, Minnesota
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Mark H Zangmeister Center - SCRI - PPDS, Columbus, Ohio
  - Tennessee Oncology NASH - SCRI - PPDS, Nashville, Tennessee
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Medical Oncology Associates - Spokane, Spokane, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Canberra Region Cancer Centre, Garran, Australia Capital Territory
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (10):
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt, Carinthia
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Ordensklinikum Linz, Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H, Linz, Upper Austria
  - Pyhrn-Eisenwurzen Klinikum Steyr, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Landeskrankenhaus Feldkirch, Rankweil, Vorarlberg
  - Kepler Universitätsklinikum Linz, Linz
  - Salzburg Cancer Research Institute, Salzburg
  - A.ö. Krankenhaus der Barmherzigen Brüder, Wein
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (11):
  - Imelda VZW, Bonheiden, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Belgique
  - Hôpital de Jolimont, La Louvière, Hainaut
  - Centre Hospitalier de l'Ardenne, Libramont, Luxembourg
  - CHU UCL Namur asbl - Site Godinne, Yvoir, Namur
  - Onze-Lieve-Vrouwziekenhuis, Aalst, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Grand Hopital de Charleroi asbl, Charleroi
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- France (5):
  - Hopitaux de La Timone, Marseille, Bouches-du-Rhône
  - Centre François Baclesse, Caen, Calvados
  - Hopital Jean Minjoz, Besançon, Doubs
  - Hôpital de Rangueil, Toulouse, Haute-Garonne
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes, Ille-et-Vilaine
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Tübingen, Tübingen
  - Klinikum Weiden, Weiden
- Italy (10):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l - PPDS, Meldola, Emilia-Romagna
  - Azienda Unita Sanita Locale di Reggio Emilia IRCCS, Reggio Emilia, Emilia-Romagna
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Instituto Europeo Di Oncologia, Milan, Lombardy
  - Ospedale degli Infermi, Candiolo, Piedmont
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Ospedale Santa Maria Della Misericordia Di Perugia, Terni, Umbria
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Venito
  - Fondazione IRCCS Policlinico San Matteo di Pavia-Vialle Camillo Golgi 19, Pavia
- South Korea (6):
  - National Cancer Center, Seoul, Gyeonggido
  - CHA Bundang Medical Center, CHA University, Seoul, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System - PPDS, Seoul, Seoul Teugbyeolsi
  - Chonnam National University Hwasun Hospital, Hwasun
  - Asan Medical Center - PPDS, Seoul
- Spain (23):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Jaen, Jaén, Jaen
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid, Madrid, Communidad Delaware
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Institut Catala d'Oncologia Girona, Girona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Center Madrid - España, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (3):
  - Aberdeen Royal Infirmary - PPDS, Aberdeen, Aberdeen City
  - Hammersmith Hospital, London, City of London
  - Derriford Hospital, Plympton, Devon

IPD SHARING:
Plan to Share IPD: No